CLINICAL TRIAL: NCT03607331
Title: Auricular Concha Electro-acupuncture for the Treatment of Mild to Moderate Depression: A Randomized Controlled Trial
Brief Title: Auricular Concha Electro-acupuncture for the Treatment of Depression
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Peijing Rong, The deputy director of Institute of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChinaACMS-5
Record Dates: First submitted 2018-05-15; First posted 2018-07-31 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Depression; Depressive Symptom; Depressive Disorder
Keywords: depression; electro-acupuncture; auricular concha
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Citalopram

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular vagus nerve stimulation (Experimental): Auricular Concha Electro-acupuncture: twice a day at home as required, once in the morning and once in the evening, with 5 consecutive days per week for two months
  Interventions: Device: Auricular vagus nerve stimulation
- Citalopram (Active Comparator): citalopram for oral administration; 10mg for the first 1-3 days, 20mg for the following 4-7 days；40mg for the left days within two months
  Interventions: Drug: Citalopram

INTERVENTIONS:
Device: Auricular vagus nerve stimulation — Auricular vagus nerve stimulation is a typical representative of TCM modernization.
  Other Names: vagus nerve stimulation at auricular concha
  Arms: Auricular vagus nerve stimulation
Drug: Citalopram — Citalopram is an antidepressant drug of the selective serotonin reuptake inhibitor (SSRI) class.It has U.S. Food and Drug Administration approval to treat major depression.
  Other Names: brand name：Cipramil, SFDA J20130028
  Arms: Citalopram

SUMMARY:
The objective of this study was to compare the therapeutic effects of Auricular Concha Electro-acupuncture and Citalopram on patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
In this study, 106 patients with MDD were randomly divided into the auricular concha electro-acupuncture group and the citalopram group by the evaluation blind method and randomized control design, and were treated for 8 weeks and 4 weeks follow-up. In No. 0, 2, 4, 6, 8, 10, 12 Weekend, Hamilton Rating Scale for Depression-17 Item (HAM-D17) and Hamilton Anxiety Rating Scale (Ham-A) were performed for all patients. During the No. 0/8 weekend, patients were tested and analyzed for peripheral blood NE, 5-HT, DA, Cortisol, ACTH, GABA, glutamic acid, BDNF and BFGF, and the brain is also examined and analyzed by fMRI.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis is consistent with DSM-V diagnostic criteria for mild-to- moderate depression;
2. Patients with the first onset or recurrence of the disease have not been treated with antidepressant or without antidepressant treatment before treatment for 3 months;
3. Age from 18 to 65 years old, with no gender;
4. Outpatient;
5. 17 Item Hamilton Depression Rating Scale (HAMD-17) score > 7, and <24;
6. Signed informed consent.

Exclusion Criteria:

1. In addition to depression, it conforms to the diagnostic criteria of any psychiatric disease;
2. Patients with a history of schizophrenia or other mental illness;
3. Patients with cognitive impairment or personality disorder;
4. In the past 6 months, patients who have met the DSM-V criteria for substance related and addictive disorders;
5. Before entering the group, any other antidepressant treatment is being accepted;
6. Patients with serious body disease, such as heart disease (namely Ⅱ and Ⅱ above cardiac function) , obvious abnormalities of liver and kidney function (Biomarkers more than 3 times normal);
7. Serious suicidal ideation or suicidal behavior.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 106 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
17 Item Hamilton Depression Rating Scale (HAMD-17) Score Change | Baseline and 1 week,baseline and 2th weeks,baseline and 4th weeks,baseline and 6th weeks,baseline and 8th weeks, baseline and 10th weeks after treatment, baseline and 12th weeks after treatment
  The Hamilton Depression Rating Scale has proven useful for determining the level of depression before, during, and after treatment. It is based on the clinician's interview with the patient and probes symptoms such as depressed mood, guilty feelings, suicide, sleep disturbances, anxiety levels and weight loss. The interview and scoring takes about 15 minutes. The rater enters a number for each symptom construct that ranges from 0 (not present) to 4 (extreme symptoms). The higher the total score is, the worse it is.The total score of 17HAMD more than 24 is defined as major depression, more than 17 but less than 24 is mild or moderate depression, and less than 7 is no depression.

SECONDARY OUTCOMES:
14 Item Hamilton Anxiety Scale (HAMA-14) Score Change | Baseline and 1 week,baseline and 2th weeks,baseline and 4th weeks,baseline and 6th weeks,baseline and 8th weeks, baseline and 10th weeks after treatment, baseline and 12th weeks after treatment
  This widely-used interview scale measures the severity of a patient's anxiety, based on 14 parameters, including anxious mood, tension, fears, insomnia, somatic complaints and behavior at the interview. The higher the total score is, the worse it is. The total score of HAMA-14 more than 29 is defined as severe anxiety, more than 21 but less than 29 is obvious anxiety, more than 14 but less than 21 is certain anxiety, more than 7 but less than 14 is likely to be anxiety, and less than 6 is no anxiety.
NE(ng/L) | Baseline and 8th week
  Biochemical indicators of peripheral blood
5-HT(ng/L) | Baseline and 8th week
  Biochemical indicators of peripheral blood
DA(ng/L) | Baseline and 8th week
  Biochemical indicators of peripheral blood
Cortisol(ng/L) | Baseline and 8th week
  Biochemical indicators of peripheral blood
ACTH(ng/L) | Baseline and 8th week
  Biochemical indicators of peripheral blood
GABA(ng/L) | Baseline and 8th week
  Biochemical indicators of peripheral blood
Glutamate(ng/L) | Baseline and 8th week
  Biochemical indicators of peripheral blood
BDNF(ng/L) | Baseline and 8th week
  Biochemical indicators of peripheral blood
bFGF(ng/L) | Baseline and 8th week
  Biochemical indicators of peripheral blood

OTHER OUTCOMES:
systolic blood pressure (mmHg) | Baseline and 8th week
  Physiological indicators
diastolic blood pressure (mmHg) | Baseline and 8th week
  Physiological indicators
respiration rate(breaths/min) | Baseline and 8th week
  Physiological indicators
pulse rate (beats/min) | Baseline and 8th week
  Physiological indicators

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Acupuncture and Moxibustion, Beijing, Beijing Municipality, China